CLINICAL TRIAL: NCT04596033
Title: A Phase 1 Study to Evaluate the Safety, Proliferation and Persistence of GEN-011, an Autologous Adoptive Cell Therapy Targeting Neoantigens in Solid Tumors
Brief Title: TiTAN-1: Safety, Proliferation and Persistence of GEN-011 Autologous Cell Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-011-101
Record Dates: First submitted 2020-09-30; First posted 2020-10-22 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma; Renal Cell Carcinoma; Small-cell Lung Cancer; Cutaneous Squamous Cell Carcinoma; Anal Squamous Cell Carcinoma; Merkel Cell Carcinoma
Keywords: Personalized; Immunotherapy; Solid Tumor; Personal; Cell Therapy; Carcinoma; Melanoma; Lung; Bladder; Cancer; Kidney; Anal; Squamous; TiTAN; ATLAS; PLANET; TiTAN-1; Autologous; Neoantigen
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Anus Neoplasms; Carcinoma, Merkel Cell; Carcinoma; Neoplasms | interventions — Interleukin-2; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multiple Low Dose (MLD) (Experimental): GEN-011 is administered by IV infusion at 4-week intervals, up to 5 doses maximum. Each dose is followed by IL-2 administration. MLD patients will not undergo lymphodepletion.
  Interventions: Biological: GEN-011; Drug: IL-2
- Single High Dose (SHD) (Experimental): GEN-011 is administered as a single IV infusion at the maximum available cell yield, after the patient completes a fludarabine/cyclophosphamide lymphodepletion regimen. The single GEN-011 dose is followed by IL-2 administration.
  Interventions: Biological: GEN-011; Drug: IL-2; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: GEN-011 — Personalized neoantigen adoptive cell therapy (ACT)
Drug: IL-2 — Cytokine
  Other Names: Interleukin-2
Drug: Fludarabine — Lymphodepletion drug
  Arms: Single High Dose (SHD)
Drug: Cyclophosphamide — Lymphodepletion drug
  Arms: Single High Dose (SHD)

SUMMARY:
TiTAN-1 is a first-in-human study of GEN-011, an experimental treatment being evaluated in adult patients with advanced cancer. GEN-011 is a T cell therapy made specific to each patient, using the patient's own circulating immune cells. First, Genocea confirms which cancer proteins are recognized already by each patient's T cells using ATLAS™. Then, immune cells that recognize these cancer proteins are multiplied many times (a process called PLANET™) to create a personalized GEN-011 cell therapy, which is given back to the patient in one or more intravenous (IV) infusions.

DETAILED DESCRIPTION:
TiTAN-1 is an open-label, multicenter, first-in-human Phase 1 study of GEN-011 in patients with melanoma, non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial carcinoma (UC, bladder, ureter, urethra, or renal pelvis), renal cell carcinoma (RCC), small cell lung cancer (SCLC), cutaneous squamous cell carcinoma (CSCC), or anal squamous cell carcinoma (ASCC). Patients will be enrolled into one of 2 cohorts. One cohort will receive a multiple low dose (MLD) regimen of GEN-011 to be given without lymphodepletion, and a second cohort will receive a single high dose (SHD) regimen of GEN-011 after lymphodepletion. Regardless of cohort, each dose of GEN-011 will be followed by a course of interleukin-2 (IL-2) as costimulatory therapy.

GEN-011 is an investigational, personalized neoantigen adoptive cell therapy (ACT) that is being developed by Genocea for the treatment of adult patients with advanced solid tumors. A proprietary tool developed by Genocea called ATLAS™ (Antigen Lead Acquisition System) will be used to identify true immunogenic neoantigens from each patient's tumor that are recognized by their own CD4 and/or CD8 T cells. ATLAS-identified neoantigens will be used to stimulate and select autologous T cells collected by apheresis to generate an adoptive cell product ex vivo.

ELIGIBILITY:
Inclusion Criteria:

* Consents to study procedures
* Diagnosis of one of the following solid tumors: cutaneous melanoma, non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial carcinoma (UC), renal cell carcinoma (RCC), small cell lung cancer (SCLC), cutaneous squamous cell carcinoma (CSCC), anal squamous cell carcinoma (ASCC), merkel cell carcinoma (MCC).
* Received, been intolerant of, or been ineligible to receive standard of care treatment regimen.
* Measurable disease per RECIST criteria
* Life expectancy > 6 months and ECOG status 0 or 1
* Capacity to tolerate lymphodepletion (SHD group only) and IL-2 therapy
* Tumor tissue available
* Willing to use contraceptives for 90 days after receiving GEN-011, and not currently pregnant.
* Adequate blood, liver, kidney, and lung function
* Sufficient stimulatory neoantigens identified in ATLAS

Exclusion Criteria:

* Receiving immunosuppressive medications
* Serious ongoing viral, bacterial, or fungal infection
* History of cardiac arrhythmias or significant heart block
* History of leptomeningeal carcinomatosis
* Active autoimmune disease
* Portal vein thrombosis
* Malignant disease other than those treated in this study
* Receiving other investigational anti-cancer therapy
* Prior stem cell or solid organ transplant
* Primary immune deficiency disease
* Significant ongoing toxicities from prior therapies
* A history of allergic reaction to sulfur derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years after first GEN-011 infusion
  Adverse events will be graded according to the NC Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
T cell responses to GEN-011 | 2 years after first GEN-011 infusion
  Antigen-specific immunogenicity assays
Duration of response | 2 years after first GEN-011 infusion
  Measured by RECIST
Progression-free survival | 2 years after first GEN-011 infusion
  Length of time without disease progression
Overall survival | From first GEN-011 infusion through study completion, at least 2 years
  Length of time patient remains alive

OTHER OUTCOMES:
Immune cell phenotyping | 2 years after first GEN-011 infusion
  Classification of peripheral immune cells via flow cytometry
Epitope Spread | 4 weeks after first GEN-011 infusion
  Tumor mutations will be identified by gene sequencing at multiple timepoints, and comparing the differences in mutations over time
Tumor infiltrating immune cell | 2 years after first GEN-011 infusion
  Quantitation and phenotyping of immune cells in proximity to tumor cells using immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Davis, MD, Study Director — Genocea Biosciences, Inc.
Locations (8):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas